CLINICAL TRIAL: NCT05489965
Title: Gender Disparities in Voice Outcomes After Tracheoesophageal Puncture in Total Laryngectomy
Brief Title: Gender Disparities in Voice Outcomes After Tracheoesophageal Puncture in Total Laryngectomy Patients (UC Davis)
Status: Recruiting | Type: Observational
Sponsor: University of California, Davis (Other)
Collaborators: University of California, San Diego (Other)
Responsible Party: Sponsor
Other Study IDs: 1509981
Record Dates: First submitted 2022-07-28; First posted 2022-08-05 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Speech Disorders; Speech Dysfunction; Laryngectomy; Status; Tracheoesophageal Prosthesis; Total Laryngectomy
MeSH Terms: conditions — Speech Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To perform a multi-site prospective study assessing, both subjectively and objectively, the gender disparities in speech outcomes of patients using TEP after total laryngectomy.

The investigators hypothesize that speech outcomes, both subjective and objective measures, will be significantly poorer for female patients compared to male patients. The outcome of the study is to prospectively assess both subjective and objective gender disparities in voice and speech outcomes of patients using TEP after total laryngectomy across a multiple institutions. The investigators hypothesize that both subjective and objective measurements of voice, speech and quality of life will be poorer for female patients in comparison to male patients.

DETAILED DESCRIPTION:
Total laryngectomy (TL) is typically performed in patients with advanced laryngeal cancer as a means of removing the entire larynx and surrounding structures that have been affected by the malignancy. Following total laryngectomy, patients lose ability to produce voice. Thus, they require the use of alternative methods of to produce voice along with extensive speech rehabilitation. Currently, there are three main speech alternative options, esophageal speech, tracheoesophageal speech, and electrolarynx speech. The focus of this study will be on patients rehabilitating their speech using tracheosophgeal speech through a tracheoesophageal prosthesis (TEP). It has been shown that generally for TL patients, better voice quality and satisfaction with voice is associated with improved quality of life. Currently, speech rehabilitation outcomes are measured with a multidimensional approach, using various scales ranging from acoustic analysis, perceptual evaluation, and patient-reported outcomes. The majority of studies analyzing outcomes in total laryngectomy patients, however, is predominated by assessment of the male laryngectomee population. Historically, this has been due to the greater incidence of laryngeal cancers in males than females. Due to this, there has been minimal research investigating potential gender differences in the laryngectomy population. Of the limited data available regarding the female laryngectomee population, it has been shown that gender frequency differences seen in normal subjects are lost following total laryngectomy and the resulting tracheoesophageal voice is more similar to the normal male voice, thus females face a greater voice handicap compared to their male counterparts (Kazi, 2006; Deore, 2011). While some studies have assessed the resulting quality of life differences between the genders in the laryngectomy population (Lee, 2010), few have investigated voice outcomes using both subjective and objective scales as used in this study. The outcomes of this study will be key to understanding what metrics are potentially contributing to the voice and lifestyle dissatisfaction that prior studies have demonstrated in the female laryngectomee population. This quantifiable data will provide a way of modifying future voice rehabilitation in the female population to enable better satisfaction and minimize gender differences in voice outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects who have completed total laryngectomy and are using TEP

Exclusion Criteria:

* Subjects who have not completed total laryngectomy and are not using TEP

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — this trial is studying the disparities amongst genders (male vs. female)
Study Population: patients with advanced laryngeal cancer who have completed total laryngectomy requiring use of alternative methods to produce voice along with extensive speech rehabilitation.
Sampling Method: Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2023-05-31 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
FACT-H&N (Functional Assessment of Cancer Therapy - Head & Neck) | Through study completion; 3 years (anticipate completion by June 2025)
  Patient reported survey.
AVHI (Alaryngeal Voice Handicap Index) | Through study completion; 3 years (anticipate completion by June 2025)
  Patient reported survey.

SECONDARY OUTCOMES:
GRBAS - Grade, Roughness, Breathiness, Asthenia, and Strain | Through study completion; 3 years (anticipate completion by June 2025)
  Examiner-based interpretation of roughness/breathiness of patient's voice. Scale of 0-3, 3 indicating severe, 0 indicating normal
Sustained phonation time | Through study completion; 3 years (anticipate completion by June 2025)
  A measurement in seconds of how long a patient can sustain phonation.
Fundamental frequency | Through study completion; 3 years (anticipate completion by June 2025)
  A measurement of frequency of voice during alaryngeal speech/sustained phonation

CONTACTS AND LOCATIONS:
Locations (1):
- University of California San Diego, La Jolla, California, United States